CLINICAL TRIAL: NCT00742872
Title: A Prospective Double-Blind Placebo-Controlled Trial of Mosapride in Patients With Constipation-Predominant Irritable Bowel Syndrome
Brief Title: Randomized Trial of Mosapride Versus Placebo in the Treatment of Constipation-Predominant Irritable Bowel Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment, high drop out rate
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Nabil Mansour, assistant professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUB-IM.AS1.21
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-02

CONDITIONS: Constipation-Predominant Irritable Bowel Syndrome
Keywords: Mosapride; Irritable Bowel Syndrome; Constipation
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Mosapride
  Interventions: Drug: Mosapride Citrate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mosapride Citrate — One 5 mg tablet taken orally three times per day (15 min before meals) for 8 weeks.
  Other Names: Mosar
  Arms: 1
Drug: Placebo — One tablet (identical in shape and form to the actual drug) taken orally three times per day (15 min before meals) for 8 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Mosapride, an agent which acts on serotonin receptors in the gastrointestinal tract, is effective in the treatment of constipation-predominant irritable bowel syndrome (C-IBS).

ELIGIBILITY:
Inclusion Criteria:

* Rome III Criteria for IBS:

Patients must have recurrent abdominal pain or discomfort at least 3 days per month during the previous 3 months that is associated with 2 or more of the following:

* Relieved by defecation
* Onset associated with a change in stool frequency
* Onset associated with a change in stool form or appearance

In addition, patients have to experience at least two of the following symptoms for at least 25% of the time [11]:

* Altered stool frequency (< 3 bowel movements per week)
* Altered stool form (lumpy/hard i.e. Bristol type I-III [see appendix 1])
* Altered stool passage (straining, urgency, or a feeling of incomplete evacuation)
* Passage of mucus, bloating, or a feeling of abdominal distension

Exclusion Criteria:

* Previous allergy to mosapride
* Nocturnal Symptoms (pain in the middle of the night, or other nocturnal symptoms which suggest an organic disease)
* Age < 18 years
* History of bloody stools or melena
* Diarrhea (>3 bowel movements per day)
* Constitutional symptoms (fever, weight loss)
* Severe constipation (< 1 bm/week)
* Pregnancy or lactation
* Patients with history of cardiac arrhythmias
* QT prolongation on baseline ECG
* Chronic laxative use and dependence
* Patients with previous history of congenital heart disease
* Patients with previous history of hypokalemia or hyperkalemia
* Patients taking the following classes of drugs: HIV antivirals, macrolides, anti-arrhythmics, and azole drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ala' I. Sharara, MD, Principal Investigator — American University of Beirut Medical Center; Nabil M. Mansour, MD, Study Director — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

RESULTS

PARTICIPANT FLOW:
Groups:
- Study: Mosapride
  Mosapride Citrate : One 5 mg tablet taken orally three times per day (15 min before meals) for 8 weeks.
- Placebo: Placebo
  Placebo : One tablet (identical in shape and form to the actual drug) taken orally three times per day (15 min before meals) for 8 weeks.
Period: Overall Study
Arm/Group | Study | Placebo
Started | 21 | 20
Completed | 9 | 12
Not Completed | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (17) | 41 (16) | 43 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Lebanon | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Adequate Relief of Symptoms Associated With Constipation-predominant Irritable Bowel Syndrome.
Time Frame: Within the first 8 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Study | Placebo
Number analyzed (Participants) | 21 | 20
participants | 7 | 10

ADVERSE EVENTS:
Arm/Group | Study | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
High placebo response rate, high dropout rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No